CLINICAL TRIAL: NCT03616106
Title: Information Visualizations to Facilitate Patient-provider Communication in HIV Care: Info Viz HIV
Brief Title: Information Visualizations to Facilitate HIV-related Patient-provider Communication (Info Viz: HIV)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Associate Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAR9023; 1K99NR017829-01A1 (NIH)
Record Dates: First submitted 2018-07-23; First posted 2018-08-06 (Actual); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Health Communication
Keywords: Information Visualization

STUDY DESIGN:
Intervention Model Description: This study will use a single group pretest-posttest design to evaluate if using infographics during clinic visits can lead to improved patient outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants in the intervention group will receive health education using infographics (Infographic Intervention) during their regularly scheduled clinic visits.
  Interventions: Other: Infographic intervention

INTERVENTIONS:
Other: Infographic intervention — All study participants will receive health education using infographics during their regularly scheduled clinic appointments.

SUMMARY:
To complete the study aims, a mixed methods study that includes a single group pretest-posttest study design will be used to pilot test the infographic intervention. In-depth interviews will be completed with a selection of participants to explore participant perceptions of HIV-related communication using infographics. Data will be collected from participants through baseline (at enrollment) and follow up assessments (at 3-, 6-, and 9-month follow up visits). Follow up interviews will be conducted with the providers involved in the intervention to ascertain their perspectives on the clinical utility of infographics.

DETAILED DESCRIPTION:
The Caribbean has among the highest HIV prevalence in the world. Regionally, the majority of HIV/AIDS cases are located on the island of Hispaniola, comprised of the Dominican Republic (DR) and Haiti. Due to a large international response and widespread availability of antiretroviral therapy (ART), in recent years the incidence of HIV in the DR has declined and prevalence hovers around 1% in the general population. The effective and long-term management of this condition depends on infected individuals being able to acquire ART and apply the learned information and self-management skills that lead to optimal adherence.

HIV-related disparities exist in developing countries, such as the DR, where minority groups and/or those with low socioeconomic status experience higher disease burdens and worse health outcomes than those with higher socioeconomic status. These disparities may be exacerbated when individuals are unable to understand the health information, as low health literacy has been associated with worse health outcomes, less use of healthcare services, poorer knowledge of illness, and worse self-management. The effective management of HIV requires patients to acquire, comprehend, and use large amounts of complex information, including how to manage variations in health status, medications and their side effects, nutrition and exercise needs, and healthy coping. Health care providers can help patients understand pertinent health information by offering it in targeted, culturally-, language-, and literacy-appropriate ways.

One such strategy is to use infographics to assist communication through visual representations of information. Participatory design of infographics supports presentation of information in a culturally appropriate and visually appealing format which can improve information understanding, health behaviors, attention span, and ability to recall information. It is critical to develop and test methods to improve the way health information is delivered to patients in these clinical contexts so patients, including those with low health literacy, can acquire and comprehend the information needed to improve self-management behavior and treatment outcomes.

Preliminary studies showed many persons living with HIV (PLWH) attending Clínica de Familia La Romana do not fully comprehend and use the health information they receive through current modalities. In response, culturally relevant, evidence-based infographics to improve information delivery during clinical visits were developed with a participatory design methodology (manuscript under review). The next phase of this study is to rigorously assess if using these infographics is a feasible, acceptable, and efficacious method to enhance HIV-related clinician-patient communication and lead to improved patient outcomes. Additionally, a thorough exploration into the cultural factors of patient-provider communication in the Dominican Republic that can influence infographic use for clinician-patient communication in a clinical setting is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥) 18 years of age
* Spanish-speaking
* Living with HIV and have a detectable viral load
* Attend Clínica de Familia La Romana
* Plan to receive care at the same clinic for the next year

Exclusion Criteria:

* Does not meet inclusion criteria
* Not able to understand study procedures or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, RN, Principal Investigator — Columbia University; Samantha B Stonbraker, PhD, MPH, RN, Study Director — Columbia University
Locations (1):
- Clínica de Familia La Romana, La Romana, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of individual participant data will be made available to qualified researchers seeking to replicate methods or to those working on a new study who need the evidence-base to do so in a rigorous way. All de-identified participant data will be shared with other researchers. Please note that all of this data will be in Spanish.
Supporting Information: CSR, Analytic Code
Time Frame: Data will be available 3 months after the publication of primary results.
Access Criteria: To request data please email the study director listed on this record with the reason you need the data and your planned use of it.

REFERENCES:
- [Background] Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, Kindelan JM, Carmona A, Juega J, Ocampo A; GEEMA Study Group. Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. AIDS. 2002 Mar 8;16(4):605-13. doi: 10.1097/00002030-200203080-00012. PMID 11873004
- [Background] Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014 Nov;67(11):1265-73. doi: 10.1016/j.jclinepi.2014.06.009. Epub 2014 Aug 3. PMID 25091546
- [Background] Bakken S, Holzemer WL, Brown MA, Powell-Cope GM, Turner JG, Inouye J, Nokes KM, Corless IB. Relationships between perception of engagement with health care provider and demographic characteristics, health status, and adherence to therapeutic regimen in persons with HIV/AIDS. AIDS Patient Care STDS. 2000 Apr;14(4):189-97. doi: 10.1089/108729100317795. PMID 10806637
- [Background] Dang BN, Westbrook RA, Hartman CM, Giordano TP. Retaining HIV Patients in Care: The Role of Initial Patient Care Experiences. AIDS Behav. 2016 Oct;20(10):2477-2487. doi: 10.1007/s10461-016-1340-y. PMID 26910339
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] De Boni R, Veloso VG, Grinsztejn B. Epidemiology of HIV in Latin America and the Caribbean. Curr Opin HIV AIDS. 2014 Mar;9(2):192-8. doi: 10.1097/COH.0000000000000031. PMID 24356327
- [Background] Figueroa JP. Review of HIV in the Caribbean: significant progress and outstanding challenges. Curr HIV/AIDS Rep. 2014 Jun;11(2):158-67. doi: 10.1007/s11904-014-0199-7. PMID 24623473
- [Background] Rojas P, Malow R, Ruffin B, Rothe EM, Rosenberg R. The HIV/AIDS Epidemic in the Dominican Republic: Key Contributing Factors. J Int Assoc Physicians AIDS Care (Chic). 2011 Sep-Oct;10(5):306-15. doi: 10.1177/1545109710397770. Epub 2011 Mar 2. PMID 21368008
- [Background] Gebre Y, Forbes NM, Peters A. Review of HIV treatment progress, gaps, and challenges in the Caribbean, 2005-2015. Rev Panam Salud Publica. 2016 Dec;40(6):468-473. PMID 28718497
- [Background] Perez-Escamilla R. Acculturation, nutrition, and health disparities in Latinos. Am J Clin Nutr. 2011 May;93(5):1163S-7S. doi: 10.3945/ajcn.110.003467. Epub 2011 Mar 2. PMID 21367946
- [Background] Barreto SM, Miranda JJ, Figueroa JP, Schmidt MI, Munoz S, Kuri-Morales PP, Silva JB Jr. Epidemiology in Latin America and the Caribbean: current situation and challenges. Int J Epidemiol. 2012 Apr;41(2):557-71. doi: 10.1093/ije/dys017. Epub 2012 Mar 9. PMID 22407860
- [Background] Wawrzyniak AJ, Ownby RL, McCoy K, Waldrop-Valverde D. Health literacy: impact on the health of HIV-infected individuals. Curr HIV/AIDS Rep. 2013 Dec;10(4):295-304. doi: 10.1007/s11904-013-0178-4. PMID 24222474
- [Background] Laws MB, Lee Y, Rogers WH, Beach MC, Saha S, Korthuis PT, Sharp V, Cohn J, Moore R, Wilson IB. Provider-patient communication about adherence to anti-retroviral regimens differs by patient race and ethnicity. AIDS Behav. 2014 Jul;18(7):1279-87. doi: 10.1007/s10461-014-0697-z. PMID 24464408
- [Background] Kalichman SC, Rompa D. Functional health literacy is associated with health status and health-related knowledge in people living with HIV-AIDS. J Acquir Immune Defic Syndr. 2000 Dec 1;25(4):337-44. doi: 10.1097/00042560-200012010-00007. PMID 11114834
- [Background] Zhang NJ, Terry A, McHorney CA. Impact of health literacy on medication adherence: a systematic review and meta-analysis. Ann Pharmacother. 2014 Jun;48(6):741-51. doi: 10.1177/1060028014526562. Epub 2014 Mar 11. PMID 24619949
- [Background] Mackey LM, Doody C, Werner EL, Fullen B. Self-Management Skills in Chronic Disease Management: What Role Does Health Literacy Have? Med Decis Making. 2016 Aug;36(6):741-59. doi: 10.1177/0272989X16638330. Epub 2016 Apr 6. PMID 27053527
- [Background] Schulman-Green D, Jaser S, Martin F, Alonzo A, Grey M, McCorkle R, Redeker NS, Reynolds N, Whittemore R. Processes of self-management in chronic illness. J Nurs Scholarsh. 2012 Jun;44(2):136-44. doi: 10.1111/j.1547-5069.2012.01444.x. Epub 2012 May 2. PMID 22551013
- [Background] Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. Self-management approaches for people with chronic conditions: a review. Patient Educ Couns. 2002 Oct-Nov;48(2):177-87. doi: 10.1016/s0738-3991(02)00032-0. PMID 12401421
- [Background] Garcia-Retamero R, Dhami MK. Pictures speak louder than numbers: on communicating medical risks to immigrants with limited non-native language proficiency. Health Expect. 2011 Mar;14 Suppl 1(Suppl 1):46-57. doi: 10.1111/j.1369-7625.2011.00670.x. PMID 21323820
- [Background] Houts PS, Doak CC, Doak LG, Loscalzo MJ. The role of pictures in improving health communication: a review of research on attention, comprehension, recall, and adherence. Patient Educ Couns. 2006 May;61(2):173-90. doi: 10.1016/j.pec.2005.05.004. Epub 2005 Aug 24. PMID 16122896
- [Background] Garcia-Retamero R, Okan Y, Cokely ET. Using visual aids to improve communication of risks about health: a review. ScientificWorldJournal. 2012;2012:562637. doi: 10.1100/2012/562637. Epub 2012 May 2. PMID 22629146
- [Background] Arcia A, Suero-Tejeda N, Bales ME, Merrill JA, Yoon S, Woollen J, Bakken S. Sometimes more is more: iterative participatory design of infographics for engagement of community members with varying levels of health literacy. J Am Med Inform Assoc. 2016 Jan;23(1):174-83. doi: 10.1093/jamia/ocv079. Epub 2015 Jul 13. PMID 26174865
- [Background] Rao JK, Anderson LA, Inui TS, Frankel RM. Communication interventions make a difference in conversations between physicians and patients: a systematic review of the evidence. Med Care. 2007 Apr;45(4):340-9. doi: 10.1097/01.mlr.0000254516.04961.d5. PMID 17496718
- [Background] Stonbraker S, Smaldone A, Luft H, Cushman LF, Lerebours Nadal L, Halpern M, Larson E. Associations between health literacy, HIV-related knowledge, and information behavior among persons living with HIV in the Dominican Republic. Public Health Nurs. 2018 May;35(3):166-175. doi: 10.1111/phn.12382. Epub 2017 Dec 29. PMID 29285785
- [Background] Stonbraker S, Befus M, Lerebours Nadal L, Halpern M, Larson E. Factors Associated with Health Information Seeking, Processing, and Use Among HIV Positive Adults in the Dominican Republic. AIDS Behav. 2017 Jun;21(6):1588-1600. doi: 10.1007/s10461-016-1569-5. PMID 27714522
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Lee SY, Stucky BD, Lee JY, Rozier RG, Bender DE. Short Assessment of Health Literacy-Spanish and English: a comparable test of health literacy for Spanish and English speakers. Health Serv Res. 2010 Aug;45(4):1105-20. doi: 10.1111/j.1475-6773.2010.01119.x. Epub 2010 May 24. PMID 20500222
- See also: Source of the Health Status Assessment published by the AIDS Clinical Trials Group (ACTG) Outcomes Committee — https://www.frontierscience.org/apps/cfmx/apps/common/QOLAdherenceForms/index.cfm?project=ACTG

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of interventionists
  Initially, 2 interventionists were enrolled, then one left the study and a replacement interventionist was recruited.
  Patient participant recruitment
  Initially, 50 participants were enrolled. Data was deleted for 6 participants due to a technical error. They were replaced with 6 additional patients.
Groups:
- Interventionists: Interventionists were the three health care providers who administered the infographic intervention to patient participants.
Period: Overall Study
Arm/Group | Intervention Group | Interventionists
Started | 56 | 3
Completed | 42 | 2
Not Completed | 14 | 1
Not completed — Removed by PI | 6 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 7 | 0

BASELINE CHARACTERISTICS:
Population: There were three providers who administered the infographic intervention to participants.
Groups:
- Providers: This group is comprised of the health care providers who administered the infographic intervention to patient participants.
- Intervention (Patient Participants): The intervention group is comprised of the patient participants who received the intervention during clinic visits.
- Total: Total of all reporting groups
Arm/Group | Providers | Intervention (Patient Participants) | Total
Number analyzed (Participants) | 3 | 50 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 49 | 52
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 26.7 [25 to 30] | 40.4 [21 to 70] | 39.5 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 28 | 31
  Male | 0 | 22 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 46 | 49
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 17 | 17
  White | 0 | 3 | 3
  More than one race | 3 | 29 | 32
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Dominican Republic | 3 | 50 | 53

OUTCOME MEASURES:

1. Primary Outcome: Association Between Mean CD4 Count at Baseline and 3-month Visit
Description: Association between mean CD4 count at baseline and 3-month visits.
Time Frame: Baseline and 3-month visit
Population: Only the intervention group was analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
cells/mm^3
  Baseline | 385.86 (271.53)
  3 months | 373.69 (243.26)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.859, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = -15.103, 95% CI 2-sided [-184.574 to 154.369]

2. Primary Outcome: Association Between Mean CD4 Count at Baseline and 6-month Visit
Description: Association between mean CD4 count at baseline and 6-month visits.
Time Frame: Baseline and 6-month visit
Population: Only the intervention group was analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
cells/mm^3
  Baseline | 385.86 (271.53)
  6 months | 414.41 (273.43)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.213, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = 28.243, 95% CI 2-sided [-16.694 to 73.179]

3. Primary Outcome: Association Between Mean CD4 Count at Baseline and 9-month Visit
Description: Association between mean CD4 count at baseline and 9-month visits.
Time Frame: Baseline and 9-month visit
Population: Only the intervention group was analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
cells/mm^3
  Baseline | 385.86 (271.53)
  9 months | 445.42 (279.25)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.031, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = 58.993, 95% CI 2-sided [5.713 to 112.274]

4. Primary Outcome: Association Between Mean Viral Load at Baseline and at 3-month Visits
Description: Test of association of mean viral load at baseline and at 3-month visits.
Time Frame: Baseline and 3-months
Population: Interventionists were not analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
copies/mL
  Baseline | 84,326 (238,545)
  3-months | 81,470 (240,834)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Viral load variables were log transformed for regression analyses; Test type: Other; p = 0.053, Regression, Linear — The p-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = -.0651, 95% CI 2-sided [-1.313 to 0.010]

5. Primary Outcome: Association Between Mean Viral Load at Baseline and at 6-month Visits
Description: Test of association of mean viral load at baseline and at 6-month visits.
Time Frame: Baseline and 6-months
Population: Interventionists were not analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
copies/mL
  Baseline | 84,326 (238,545)
  6-months | 91,590 (284090)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.008, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = -1.601, 95% CI 2-sided [-2.761 to -0.442]

6. Primary Outcome: Association Between Mean Viral Load at Baseline and at 9-month Visits
Description: Test of association of mean viral load at baseline and at 9-month visits.
Time Frame: Baseline and 9-months
Population: Interventionists were not analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
copies/mL
  Baseline | 84,326 (238,545)
  9-months | 45,581 (151,116)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = -2.674, 95% CI 2-sided [-3.934 to -1.415]

7. Secondary Outcome: Satisfaction With Care Scale Score
Description: 3 questions from the overall evaluation of the HIV clinic scale were administered for a total of 19 possible points on this scale. Range of possible scores is 1-19, with 19 being highest possible satisfaction with care. The breakdown of scoring by question is as follows:
  * Question 1 is a 1-7 scale with 1 being completely unsatisfied and 7 being completely satisfied
  * Question 2 is a 1-5 scale where 1 is definitely not and 5 is definitely yes
  * Question 3 is a 1-7 scale where 1 is terrible and 7 is marvelous
Time Frame: Baseline, 3-, 6-, and 9-month visits
Population: Interventionists did not receive the intervention and, therefore, are not included in the analysis of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 18.04 (1.37)
  3-months | 18.52 (0.58)
  6-months | 18.49 (0.55)
  9-months | 18.31 (0.47)

8. Secondary Outcome: Medication Adherence
Description: Adherence will be measured with the validated simplified medication adherence questionnaire (SMAQ)-6 scale, a 6-item questionnaire. A person is considered "non-adherent" if there is a "yes" answer for any of items 1,2,3, and 5. Additionally, if they answer that they have missed more than two doses in the past week (item 4) or if they have gone more than two days without taking their medication in the past 3 months (item 6). Therefore, participants are classified as either adherent or not adherent based on their answers to these questions. Any participant that didn't complete study visits or did not answer that question was considered "missing."
Time Frame: Baseline, 3-, 6-, and 9-month visits
Population: Interventionists were not exposed to the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
Participants
  Baseline: Adherent | 9
  Baseline: Non-adherent | 41
  Baseline: Missing | 0
  3-months: Adherent | 24
  3-months: Non-adherent | 22
  3-months: Missing | 4
  6-months: Adherent | 28
  6-months: Non-adherent | 15
  6-months: Missing | 7
  9-months: Adherent | 39
  9-months: Non-adherent | 3
  9-months: Missing | 8

9. Secondary Outcome: Participant's Self-reported Health-related Quality of Life Score - Physical Functioning
Description: Health-related quality of life will be measured with the Patient-Reported Outcomes Measurement Information System® (PROMIS)-29 measure, which measures 7 domains of health-related quality of life with 4 questions in each section pertaining to how that participant's health influences their life. In general, each question has five response options ranging in values from 1-5. To find the total raw score for this form with all the questions answered, the values from the responses of each question are summed. Raw scores are then translated into a T-score for each participant, which rescales the raw score into a standardized T-score with a mean of 50 and standard deviation (SD) of 10. Consequently, a person with a T-score of 40 would be one SD below the mean.
Time Frame: Up to 9 months from baseline
Population: Interventionists did not receive the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
t-score
  Baseline | 55.37 (4.20)
  3-months | 57 (0.00)
  6-months | 56.2 (3.11)
  9-months | 56.64 (2.33)

10. Secondary Outcome: Participants' Self-reported Health Status Over Past 4 Weeks.
Description: General health status was assessed with one item where participants are asked to rank their health in the past four weeks as excellent, good, fair, poor, or very poor. Results are presented as the number of participants that self-rated their health in each of those categories.
Time Frame: Baseline, 3-months, 6-months, and 9-months
Population: Interventionists did not receive the intervention and, therefore, are not included in analyses of outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
Participants
  Baseline: Excellent | 7
  Baseline: Good | 8
  Baseline: Fair | 16
  Baseline: Poor | 16
  Baseline: Very poor | 1
  Baseline: Missing | 2
  3-months: Excellent | 21
  3-months: Good | 9
  3-months: Fair | 13
  3-months: Poor | 5
  3-months: Very poor | 0
  3-months: Missing | 2
  6-months: Excellent | 13
  6-months: Good | 19
  6-months: Fair | 9
  6-months: Poor | 2
  6-months: Very poor | 0
  6-months: Missing | 7
  9-months: Excellent | 8
  9-months: Good | 21
  9-months: Fair | 13
  9-months: Poor | 0
  9-months: Very poor | 0
  9-months: Missing | 8

11. Secondary Outcome: Health Literacy
Description: Health literacy will be assessed using the short assessment of health literacy- Spanish. Scores range from 0 - 18 and above a 15 indicates that participants are likely to have adequate health literacy. Participants are then categorized as health literate or not health literate. The final number of participants who are health literate are reported here.
Time Frame: Baseline visit only
Population: Interventionists were not exposed to the intervention. Therefore, they are not included in the analyses of outcome measures.
Measure: Number; unit: Participants
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
Participants | 18

12. Secondary Outcome: Percent of Participants Who Complete an In-depth Qualitative Interview
Description: Participants will be invited to participate in an in-depth qualitative interview regarding their experiences. The number who participate will be reported as a percent of the total who are enrolled.
Time Frame: 9 months from baseline
Population: The percentage of participants who agreed to participate in an in-depth interview.
Measure: Number; unit: percent of participants
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
percent of participants | 52

13. Secondary Outcome: Participant's Self-reported Health-related Quality of Life Score - Anxiety
Description: as for outcome 9
Time Frame: Baseline, 3-, 6-, and 9-months
Population: Interventionists did not receive the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
t-score
  Baseline | 54.09 (11.54)
  3-months | 44.33 (8.18)
  6-months | 46.23 (9.45)
  9-months | 42.5 (6.92)

14. Secondary Outcome: Participant's Self-reported Health-related Quality of Life Score - Depression
Description: as for outcome 9
Time Frame: Baseline, 3-, 6-, and 9-months
Population: Interventionists did not receive the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
t-score
  Baseline | 53.40 (11.49)
  3-months | 45.51 (8.64)
  6-months | 45.27 (8.02)
  9-months | 43.19 (6.9)

15. Secondary Outcome: Participant's Self-reported Health-related Quality of Life Score - Fatigue
Description: as for outcome 9
Time Frame: Baseline, 3-, 6-, and 9-months
Population: Interventionists did not receive the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
t-score
  Baseline | 42.46 (10.01)
  3-months | 38.06 (8.01)
  6-months | 36.38 (5.65)
  9-months | 34.76 (3.88)

16. Secondary Outcome: Participant's Self-reported Health-related Quality of Life Score - Sleep Disturbance
Description: as for outcome 9
Time Frame: Baseline, 3-, 6-, and 9-months
Population: Interventionists did not receive the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
t-score
  Baseline | 45.37 (12.04)
  3-months | 40.60 (8.58)
  6-months | 41.70 (5.74)
  9-months | 43.54 (6.31)

17. Secondary Outcome: Participant's Self-reported Health-related Quality of Life Score - Social Activity Participation
Description: as for outcome 9
Time Frame: Baseline, 3-, 6-, and 9-months
Population: Interventionists did not receive the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
t-score
  Baseline | 60.91 (6.98)
  3-months | 63.65 (2.84)
  6-months | 63.83 (2.46)
  9-months | 63.72 (3.09)

18. Secondary Outcome: Participant's Self-reported Health-related Quality of Life Score - Pain Interference
Description: as for outcome 9
Time Frame: Baseline, 3-, 6-, and 9-months
Population: Interventionists did not receive the intervention and are, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
t-score
  Baseline | 46.11 (7.08)
  3-months | 42.52 (3.19)
  6-months | 42.88 (3.64)
  9-months | 43.59 (5.10)

19. Secondary Outcome: Satisfaction With Provider Scale Score at Each Time Point
Description: 4 questions from the overall evaluation of the health care provider scale were administered for a total score of 29. The range of scores is 3-29, with 29 being the highest possible satisfaction with their health care provider. The scoring breakdown by each included question is as follows:
  * Question 1 is 1- 7 points where 1 is completely dissatisfied and 7 is completely satisfied
  * Question 2 is providing an integer value of trust in care provider on a scale from 1 to 10
  * Question 3 is 1- 7 points where 1 is terrible and 7 is marvelous
  * Question 4 is 0- 5 points where 0 is definitely not and 5 is definitely yes
Time Frame: Baseline, 3-, 6-, and 9-month visits
Population: Interventionists did not receive the intervention and, therefore, are not included in the analysis of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 26.96 (3.25)
  3-months | 27.69 (1.39)
  6-months | 27.49 (1.56)
  9-months | 27.64 (1.01)

20. Secondary Outcome: Association Between Mean HIV-related Knowledge Scores at Baseline and 3-month Visits.
Description: 14 questions pertaining to HIV-related knowledge were developed according to the information that will be included in the intervention. Participants will receive one point for each correct answer and then the scores for each question will be summed to obtain a final score. Therefore, the minimum score will be 0 and maximum score will be 14 where the scores closer to 14 indicate patients have more HIV-related knowledge.
Time Frame: Baseline and 3-month visits
Population: Interventionists were not included in the assessment of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 10.26 (2.4)
  3-months | 12.43 (1.53)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = 2.172, 95% CI 2-sided [1.448 to 2.895]

21. Secondary Outcome: Association Between Mean HIV-related Knowledge Scores at Baseline and 6-month Visits.
Description: as for outcome 20
Time Frame: Baseline and 6-month visits
Population: Interventionists were not included in the assessment of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 10.26 (2.4)
  6-months | 13.14 (1.39)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = 2.872, 95% CI 2-sided [2.100 to 3.643]

22. Secondary Outcome: Association Between Mean HIV-related Knowledge Scores at Baseline and 9-month Visits.
Description: as for outcome 20
Time Frame: Baseline and 9-month visits
Population: Interventionists were not included in the assessment of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 10.26 (2.4)
  9-months | 13.44 (0.68)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Regression, Linear — This p-value is not adjusted for multiple comparisons and the a priori threshold for statistical significance was 0.05; Slope = 3.166, 95% CI 2-sided [2.487 to 3.846]

23. Secondary Outcome: Association of Engagement With Clinician Scale Score at Baseline and 3-months.
Description: The Engagement with Health Care Providers scale is a 13 item scale through which clients rate how they feel about their interactions with their providers. Answers are recorded on a 4-point scale (1=always true and 4=never true). The range of scores is between 13 and 52. Lower scores (with 13 being the lowest score) indicate more provider engagement.
Time Frame: Baseline and 3-months
Population: Interventionists did not receive the intervention and were, therefore, not included in outcome measure analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 13 [13 to 16]
  3-months | 13 [13 to 13]
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.0011, Wilcoxon signed rank — The p-value was adjusted for multiple comparisons using the Bonferroni correction. Therefore, the threshold for statistical significance was p≤0.05/3 = .017. Please see statistical analysis plan for further details; Z Score = 3.25

24. Secondary Outcome: Association of Engagement With Clinician Scale Score at Baseline and 6-months.
Description: as for outcome 23
Time Frame: Baseline and 6-months
Population: Interventionists did not receive the intervention and were, therefore, not included in outcome measure analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 13 [13 to 16]
  6-months | 13 [13 to 13]
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.0001, Wilcoxon signed rank — [p-value comment as in outcome 23, analysis 1]; Z score = 3.94

25. Secondary Outcome: Association of Engagement With Clinician Scale Score at Baseline and 9-months.
Description: as for outcome 23
Time Frame: Baseline and 9-months
Population: Interventionists did not receive the intervention and were, therefore, not included in outcome measure analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 13 [13 to 16]
  9-months | 13 [13 to 13]
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Wilcoxon signed rank — [p-value comment as in outcome 23, analysis 1]; Z score = 4.12

26. Secondary Outcome: Association Between SEMCD Scale Score at Baseline and 3-month Visits
Description: Self-efficacy to manage chronic disease scale (SEMCD) will be used. This is a 6-item measure where 1 is not at all confident and 10 is completely confident. The total range of scores is 1-10. Final scores are calculated as the mean of the 6 questions, where higher scores indicate higher self-efficacy.
Time Frame: Baseline, 3-month visits
Population: Interventionists did not receive the intervention and were, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 7.16 (2.7)
  3-months | 9.07 (1.07)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Regression, Linear — This p-value was not adjusted for multiple comparisons. The p-value threshold for statistical significance was, therefore, 0.05; Slope = 1.935, 95% CI 2-sided [1.055 to 2.815]

27. Secondary Outcome: Association Between SEMCD Scale Score at Baseline and 6-month Visits
Description: as for outcome 26
Time Frame: Baseline, 6-month visits
Population: Interventionists did not receive the intervention and were, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 7.16 (2.7)
  6-months | 9.27 (0.58)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Regression, Linear — The p-value was not adjusted for multiple comparison, therefore, the threshold for statistical significance was 0.05; Slope = 2.123, 95% CI 2-sided [1.184 to 3.062]

28. Secondary Outcome: Association Between SEMCD Scale Score at Baseline and 9-month Visits
Description: as for outcome 26
Time Frame: Baseline, 9-month visits
Population: Interventionists did not receive the intervention and were, therefore, not included in the analyses of outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
score on a scale
  Baseline | 7.16 (2.7)
  9-months | 9.7 (0.46)
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.000, Regression, Linear — The p-value was not adjusted for multiple comparison, therefore, the threshold for statistical significance was 0.05; Slope = 2.552, 95% CI 2-sided [1.612 to 3.492]

29. Secondary Outcome: Association Between Current Self-reported Health Status as Reported at Baseline and 3-months
Description: Participants are asked to rank their current health status on a scale between 0 and 100 where 0 is "death" or the worst possible health (as bad or worse than being dead) and 100 is "perfect health", or the best possible health (without HIV infection).
Time Frame: Baseline, 3-months
Population: Interventionists were not included in the intervention and were, therefore, not included in the analyses of outcome measures.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
units on a scale
  Baseline | 90 [70 to 100]
  3-months | 90 [89.5 to 100]
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.1167, Wilcoxon signed rank — The p-value was adjusted for multiple comparisons using the Bonferroni correction. Therefore, the a priori threshold for statistical significance was p≤0.05/3 = .017. For more details please see the statistical plan; Z score = -1.57

30. Secondary Outcome: Association Between Current Self-reported Health Status as Reported at Baseline and 6-months
Description: as for outcome 29
Time Frame: Baseline, 6-months
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
units on a scale
  Baseline | 90 [70 to 100]
  6-months | 95 [90 to 100]
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.0036, Wilcoxon signed rank — [p-value comment as in outcome 29, analysis 1]; Z score = -2.91

31. Secondary Outcome: Association Between Current Self-reported Health Status as Reported at Baseline and 9-months
Description: as for outcome 29
Time Frame: Baseline, 9-months
Population: as for outcome 29
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention (Patient Participants)
Number analyzed (Participants) | 50
units on a scale
  Baseline | 90 [70 to 100]
  9-months | 98 [90 to 100]
Statistical Analysis 1: Comparison: Intervention (Patient Participants); Test type: Other; p = 0.0004, Wilcoxon signed rank — [p-value comment as in outcome 29, analysis 1]; Z score = -3.54

ADVERSE EVENTS:
Time Frame: Up to 9 months
Description: Our definition of adverse event does not differ from clinicaltrials.gov definitions.
Arm/Group | Intervention Group | Interventionists
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/3
Other Adverse Events (participants affected / at risk) | 0/50 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT03616106/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03616106/SAP_001.pdf